CLINICAL TRIAL: NCT03025243
Title: The Effect of Printing Layer Thickness on the Accuracy of Computer Aided Surgical Guides : A Randomized Clinical Trial
Brief Title: The Effect of Printing Layer Thickness on the Accuracy of Computer Aided Surgical Guides
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Ahmed Hanafy, Master students, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CEBC-CU-2017-01-08
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Guided Surgery
Keywords: computer aided design , dental implants , accuracy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50 micron (Experimental): surgical guide constructed with 3D printing with printing layer thickness 50 micron
  Interventions: Device: computer aided surgical guide
- 100 micron (Active Comparator): surgical guide constructed with 3D printing with printing layer thickness 100 micron
  Interventions: Device: computer aided surgical guide

INTERVENTIONS:
Device: computer aided surgical guide — comparing accuracy of surgical guide of printing layer thickness of 50 micron and 100 micron by superimposition of pre-operative and post-operative CBCT
  Other Names: surgical guide

SUMMARY:
The purpose of this study is to evaluate the effect of printing layer thickness on accuracy of computer aided surgical guide

DETAILED DESCRIPTION:
Computer aided surgical guide has many variables that affect its accuracy , in this study one variable is considered that may affect the accuracy of surgical guide which is printing of layer thickness of surgical guide whether 50 micron or 100 micron.

computer aided surgical guide is constructed by imaging the patient pre-operative cone beam CT wearing scan appliance , then virtual implant placement on special soft ware ( Blue sky Bio ) and optical scanning of patient casts , afterword superimposition of the virtual implants on the scanned casts to design the surgical guide and printing on 3D printer ( Zenith 3D printer , Dentis , Korea ) with printing layer thickness 50 micron in first group and 100 micron in second group . Fixation of surgical guide in patient mouth and drilling of implant osteotomy through the guiding sleeves , post-operative Cone Beam CT with the same apparatus and setting as pre-operative scan .

Finally, the pre-operative and post operative scans were then overlapped to measure linear and angular deviation of the virtually planned and actual implants position.

ELIGIBILITY:
Inclusion Criteria:

* patients partially or totally edentulous arches .
* patients with Bucco-lingual bone thickness >6 mm allowing flapless implant placement
* patients free from any systemic diseases that may affect bone quality e.g diabetes .

Exclusion Criteria:

* patients with thin ridges.
* patients with systemic disease that may affect bone quality.
* Patients with poor oral hygiene and active periodontal diseases.
* Anatomical situations requiring regenerative procedure.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of surgical guide | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud El far, phd, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided